CLINICAL TRIAL: NCT06775470
Title: Impatto Delle Diverse Varianti Dei Geni BRCA1/2 su Risposta Alla Terapia e Prognosi Del Carcinoma Ovarico
Brief Title: Impact of Different BRCA1/2 Gene Variants on Response to Therapy and Prognosis of Ovarian Cancer
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: IMBARCO
Record Dates: First submitted 2024-11-28; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-10

CONDITIONS: Ovarian Cancer
Keywords: BRCA1; BRCA2; PARP
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Genes, BRCA1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Patients must have been diagnosed with ovarian cancer and be BRCA positive — Patients must have been diagnosed with ovarian carcinoma by 31/12/2021, have undergone BRCA testing at the UOC of Medical Genetics of the IRCCS AOU of Bologna Policlinico S. Orsola by 31/12/2021 and have been taken on for follow-up and/or treatment at the Medical Oncology - Zamagni and/or Gynaecological Oncology - De Iaco of the IRCCS Azienda Ospedaliero-Universitaria (AOU) of Bologna for a period of time of at least 1 year and by 31/12/2021 and for a minimum period of 6 months.
Diagnostic Test: BRCA1 and BRCA2 positive, and be affected by Ovarian Cancer — Patients must have been diagnosed with ovarian carcinoma by 31/12/2021, have undergone BRCA testing at the UOC of Medical Genetics of the IRCCS AOU of Bologna Policlinico S. Orsola by 31/12/2021 and have been taken on for follow-up and/or treatment at the Medical Oncology - Zamagni and/or Gynaecological Oncology - De Iaco of the IRCCS Azienda Ospedaliero-Universitaria (AOU) of Bologna for a period of time of at least 1 year and by 31/12/2021 and for a minimum period of 6 months.

SUMMARY:
Identify any significant differences in terms of drug response and survival between the different possible alterations in the BRCA1/2 genes, in order to stratify ovarian cancer patients with a view to increasingly personalised and thus effective therapy.

DETAILED DESCRIPTION:
Ovarian carcinoma (OC) is the leading cause of death among gynaecological neoplasms. It is, in fact, a neoplasm that is not very frequent but highly lethal: in Emilia-Romagna, the incidence is about 17 cases per 100,000 inhabitants and the mortality rate is around 15 cases per 100,000, with a very high mortality/incidence ratio (0.83). The high mortality rate is mainly due to the fact that, due to the non-specific and late symptoms, 75-80% of patients arrive at the diagnosis at an advanced stage of the disease (III-IV), characterised by a 5-year survival of less than 25%.

The primary therapeutic approach for this tumour is a combination of debulking surgery and platinum-based chemotherapy generally associated with taxanes, while as far as maintenance therapies are concerned, PARP inhibitors (PARPi), drugs capable of blocking a DNA repair mechanism alternative to that of homologous recombination, have been gaining in importance in recent years. They have proved particularly effective in tumours that present alterations in the BRCA1 and BRCA2 genes, which are key players in homologous recombination. For this reason, the detection of mutations in the BRCA1 and BRCA2 genes is predictive of the efficacy of PARPi maintenance therapy and, consequently, as of 2015, the BRCA test has been indicated in all women newly diagnosed with ovarian cancer (excluding borderline and mucinous forms), possibly from tumour tissue, given the evidence that in addition to constitutional (inherited) variants, somatic variants (acquired and tumour-confined), present in about 9%, are also associated with a PARPi benefit.

Recent data, however, have challenged the assumption that functionally significant variants for which a predisposing role has been demonstrated for hereditary breast and ovarian cancers are necessarily predictive of drug response. Furthermore, the fact that somatic mutations are present in only a limited fraction of the DNA copies analysed in a tumour suggests that there may be residual BRCA activity that compromises effective PARPi activity.

ELIGIBILITY:
Inclusion Criteria:

* ovarian cancer diagnosis by 31/12/2021;
* BRCA test at the UOC of Medical Genetics of the IRCCS AOU of Bologna Policlinico S.Orsola by 31/12/2021;
* follow-up and/or treatment at Medical Oncology and/or Gynaecological Oncology of the IRCCS Azienda Ospedaliero-Universitaria (AOU) of Bologna for a period of time of at least 1 year and by 31/12/2021 and for a minimum period of 6 months

Exclusion Criteria:

* ovarian carcinoma of 'mucinous' or 'borderline' histotype.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: From 2012 to the end of 2021, 869 patients underwent BRCA testing at the UOC of Medical Genetics of the IRCCS AOU of Bologna Policlinico S.Orsola 869 patients with CO, almost all of whom have given informed consent to the acquisition of clinical documentation relating to their case and to the use of their data for scientific purposes and about half of them were taken on for a period of at least 1 year at the Medical Oncology - Zamagni and/or the Gynaecological Oncology - De Iaco. The investigators estimated a sample of about 300 patients.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in BRCA1/2 status for predictive response to chemotherapy | 12 months
  The primary objective of the study is to clarify whether differences in the status of BRCA1/2 (presence/absence of germline and/or somatic) may be predictive in the response to chemotherapy and survival of patients with ovarian cancer.

SECONDARY OUTCOMES:
Differences in response to chemotherapy based on BRCA variant | 12 months
  The secondary objective is to determine whether among the variant carriers germline and/or somatic pathogenesis of BRCA1/2 differences exist in terms of response to chemotherapy and survival based on the specific variant found.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Turchetti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No